CLINICAL TRIAL: NCT01182831
Title: A Randomized Trial Comparing Fluoroscopy Guided Percutaneous Technique Versus Endoscopic Ultrasound Guided Technique of Celiac Plexus Neurolysis for Treatment of Pain in Carcinoma Pancreas
Brief Title: Trial Comparing Two Techniques of Celiac Plexus Neurolysis for Treatment of Pain in Carcinoma Pancreas
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Dr.Santosh Darisetty, Asian Institute of Gastroenterology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIG-GIA-201001
Record Dates: First submitted 2010-08-14; First posted 2010-08-17 (Estimated); Last update posted 2010-08-30 (Estimated); Status verified 2010-08

CONDITIONS: Pancreatic Cancer
Keywords: carcinoma pancreas; percutaneous celiac plexus neurolysis; endosonography guided celiac plexus neurolysis
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- percutaneous fluoro guided celiac plexus neurolysis (Active Comparator)
  Interventions: Procedure: percutaneous fluoro guided celiac plexus neurolysis
- EUS guided neurolysis (Active Comparator)
  Interventions: Procedure: EUS guided neurolysis

INTERVENTIONS:
Procedure: percutaneous fluoro guided celiac plexus neurolysis — It is percutaneous injection of neurolytic agent in and around the celiac ganglion
  Arms: percutaneous fluoro guided celiac plexus neurolysis
Procedure: EUS guided neurolysis — It is injection of neurolytic agent in and around the celiac ganglion using an echo endoscope.
  Arms: EUS guided neurolysis

SUMMARY:
Coeliac plexus neurolysis (CPN) is a management option for pain control in carcinoma pancreas.CPN is conventionally performed by percutaneous technique with fluoroscopic guidance. Endoscopic ultrasound (EUS) is increasingly used for CPN as it offers a better visualization of the plexus. There are limited data comparing the two modalities.The patients are on follow-up for 6 months post neurolysis.

DETAILED DESCRIPTION:
Carcinoma pancreas patients with abdominal pain requiring daily analgesics for more than 4 weeks were included.we are randomising about 100 patients into two groups to undergo either of the two procedures, i.e. celiac plexus neurolysis by percutaneous technique or by endoscopic ultrasound guided technique.The pain scores have been recorded by visual analogue scale for an average follow-up of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* all patients with carcinoma pancreas

Exclusion Criteria:

* patients below 18 years of age and who have not given consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
immediate pain relief | day of block to six months of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Andhra Pradesh, India